CLINICAL TRIAL: NCT06355895
Title: The Effect of Liver Volume Variation on Stereotactic Body Radiation Therapy (SBRT) Planning and Delivery for Upper Abdominal Malignancies
Brief Title: Liver Volume Variation Effect on SBRT Planning and Delivery for Upper Abdominal Malignancies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: American College of Radiation Oncology (Unknown)
Responsible Party: Principal Investigator, Susannah Ellsworth, Clinical Associate Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HCC 23-104
Record Dates: First submitted 2024-04-02; First posted 2024-04-10 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Upper Abdominal Malignancies
Keywords: Stereotactic Body Radiation Therapy (SBRT); Four-Dimensional Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- High Carbohydrate Diet (Experimental): 1. First scan: after an overnight fast of at least 8 hours using standard radiation oncology CT scan with contrast for treatment planning.
  2. Standardized high-carb meal such as 8 ounces of Ensure® nutritional protein shake or a similar meal, immediately following first scan and consumed within 15 minutes.
  3. Second scan: within 1 hour of ingestion of the high-carb meal using similar settings to those used in the first scan except for contrast use.
  4. Third CT scan at least 4 hours (but no more than 5 hours) after ingestion of high-carb diet on the same day utilizing same set up used in first scan with exception for the use of contrast.
  Interventions: Dietary Supplement: Standardized high-carbohydrate meal

INTERVENTIONS:
Dietary Supplement: Standardized high-carbohydrate meal — 8 ounces of Ensure® nutritional protein shake or a similar meal

SUMMARY:
Standard planning constraints for liver SBRT incorporate strict dose-volume limits for normal liver parenchyma to minimize the risk of radiation-induced liver disease. The presence of diurnal and fasting/fed variations in liver volume therefore carry substantial potential for introducing errors into estimates of dose-volume distribution within normal liver tissue, as well as affecting day-to-day setup fidelity and organ alignment for treatment. This prospective study will examine how diurnal and fast-fed variations in liver volume affect treatment planning for abdominal SBRT.

DETAILED DESCRIPTION:
Stereotactic body radiotherapy (SBRT) is an integral tool in the management of thoracic and upper abdominal malignancies. SBRT delivers ablative radiation doses in a limited number of fractions (thereby reducing interruptions in systemic therapy) with emerging evidence for feasibility and local control benefit. Effective SBRT delivery requires high-precision target localization that accounts for positional variations in both the target and nearby organs at risk (OAR). An absolute requirement for SBRT is accurate target localization and motion management, particularly when treating targets in the chest and abdomen, which are subject to respiratory motion as well as changes in configuration due to deformation of hollow viscera. To ensure adequate targeting, various technical solutions are available, including motion management approaches such as four-dimensional computed tomography (4D-CT), abdominal compression, respiratory gating, and breath hold, as well as daily image-guided radiotherapy (IGRT) techniques such as cone beam computed tomography (CBCT), which facilitate precise daily target verification and minimization of the planning target volumes (PTVs). While the effects of respiratory motion on patient positioning during upper abdominal SBRT are relatively well understood, little is known about the effect of liver volume changes on radiotherapy (RT) dose delivery, despite the potential for morphological variations in the liver to affect patient setup and radiation dose distribution in real time. The liver is a dynamic organ with various functions including glycogen storage, carbohydrate (carb)/lipid/protein metabolism, bile secretion, synthesis of plasma proteins, and metabolism of various substances including steroid hormones and ingested toxins. Liver function is affected by fasting and feeding cycles, with an intrinsic circadian rhythm first observed in animal studies. This trial proposes to affect liver volume to ultimately and positively affect treatment planning for abdominal SBRT.

ELIGIBILITY:
Inclusion Criteria:

• Have primary upper abdominal (pancreatic, bile duct, liver) cancer or upper abdominal metastases (liver, adrenal, upper abdominal lymph nodes) planned to undergo SBRT.

Exclusion Criteria:

* Had prior Radiation Therapy to the liver
* Contraindication to receipt of iodinated IV contrast for CT (such as renal insufficiency or allergy that cannot be overcome by premedication)
* Pregnancy/lactation OR woman of childbearing potential who is unable or unwilling to use adequate contraception during Radiation Therapy.
* Inability to fast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Diurnal Difference in Liver Volumes | At baseline and at 4 hours post intervention
  Percentage diurnal difference in total liver volumes (change in liver volume), as measured by Stereotactic Body Radiation Therapy (SBRT) planning software.

SECONDARY OUTCOMES:
Difference in total liver volume | At baseline and at 1 hour post intervention
  Percentage difference in total liver volume (measured by Stereotactic Body Radiation Therapy (SBRT) planning software) after standardized high-carb meal (intervention).
Percentage diurnal difference in liver mean dose at V5 Gy | At baseline and at 1 hour post intervention
  Percentage diurnal difference in liver mean dose at V5 Gy (measured by Stereotactic Body Radiation Therapy (SBRT) planning software) after standardized high-carb meal (intervention).
Percentage diurnal difference in liver mean dose at V15Gy | At baseline and at 1 hour post intervention
  Percentage diurnal difference in liver mean dose at V15 Gy (measured by Stereotactic Body Radiation Therapy (SBRT) planning software) after standardized high-carb meal (intervention).
Difference in liver mean dose at V15 Gy | At baseline and at 1 hour post intervention
  Percentage difference in liver mean dose, V5 Gy (measured by Stereotactic Body Radiation Therapy (SBRT) planning software) after standardized high-carb meal (intervention).
Difference in liver dose at V15 Gy | At baseline and at 1 hour post intervention
  Percentage difference in liver mean dose at V15 Gy (measured by Stereotactic Body Radiation Therapy (SBRT) planning software) after standardized high-carb meal (intervention).

CONTACTS AND LOCATIONS:
Overall Officials: Susannah Ellsworth, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No